CLINICAL TRIAL: NCT00422227
Title: A Randomized, Open-Label Study in the Asia-Pacific Region Comparing the Safety and Efficacy of Etanercept With Usual DMARD Therapy in Subjects With Rheumatoid Arthritis
Brief Title: Study Comparing Etanercept With Usual DMARD Therapy in Subjects With Rheumatoid Arthritis in the Asia Pacific Region
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0881A1-408
Record Dates: First submitted 2007-01-11; First posted 2007-01-15 (Estimated); Results first posted 2010-08-30 (Estimated); Last update posted 2010-08-30 (Estimated); Status verified 2010-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Methotrexate; Sulfasalazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Etanercept + Methotrexate
  Interventions: Drug: Etanercept , Methotrexate
- 2 (Active Comparator): DMARD therapy Methotrexate + Sulfasalazine/Hydroxychloroquine/Leflunomide
  Interventions: Drug: Methotrexate; sulfasalazine; hydroxychloroquine;leflunomide

INTERVENTIONS:
Drug: Etanercept , Methotrexate — * Etanercept: 25 mg twice weekly over 16 weeks, SC
  * Methotrexate: > 7.5 mg/week and no more than 25 mg/week, PO
  Arms: 1
Drug: Methotrexate; sulfasalazine; hydroxychloroquine;leflunomide — * Methotrexate: at least 7.5 mg/wk and not more than 25 mg/wk.;PO
  * Sulfasalazine: Start treatment w/500 mg daily for 1 wk, thereafter increase dose by 1 tab each wk to a max of 3 g/day;PO
  * Hydroxychloroquine:400 mg daily in divided dose, may be reduced to 200 mg. Max: 6.5 mg/kg/day
  * Leflunomide: Initially, loading dose 100 mg daily for 3 days. Maintenance: 20 mg daily
  Arms: 2

SUMMARY:
The purpose of this study is to compare the efficacy of etanercept with usual disease-modifying anti-rheumatic drug (DMARD) therapy in the treatment of moderate to severe rheumatoid arthritis (RA) over 16 weeks in the Asia Pacific region.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA
* Currently receiving an adequate dose of methotrexate (MTX) for treatment of RA
* Active RA at time of screening and baseline

Exclusion Criteria:

* Previous or current treatment with etanercept (ETN), other tumor necrosis factor-alpha inhibitors, or other biologic agents
* Concurrent treatment with a DMARD, other than MTX, at screening
* Receipt of any DMARD, other than MTX, within 3 months before screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Hong Kong: medinfo@wyeth.com; Trial Manager, Principal Investigator — For Taiwan: medinfo@wyeth.com
Locations (19):
- Hong Kong, Hong Kong
- India (3):
  - Bangalore
  - Hyderabaad
  - New Delhi
- Malaysia (5):
  - Ipoh, Perak
  - Kuala Lumpur
  - Pulau Pinang
  - Putrajaya
  - Seremban
- Philippines (4):
  - Cebu
  - Makati City
  - Manila
  - Quezon City
- Singapore, Singapore
- South Korea (2):
  - Incheon, Korea
  - Seoul, Korea
- Taiwan (2):
  - Kaohsiung City
  - Taipei
- Bangkok, Thailand

REFERENCES:
- [Derived] Fleischmann R, Koenig AS, Szumski A, Nab HW, Marshall L, Bananis E. Short-term efficacy of etanercept plus methotrexate vs combinations of disease-modifying anti-rheumatic drugs with methotrexate in established rheumatoid arthritis. Rheumatology (Oxford). 2014 Nov;53(11):1984-93. doi: 10.1093/rheumatology/keu235. Epub 2014 Jun 6. PMID 24907147
- [Derived] Bae SC, Gun SC, Mok CC, Khandker R, Nab HW, Koenig AS, Vlahos B, Pedersen R, Singh A. Improved health outcomes with etanercept versus usual DMARD therapy in an Asian population with established rheumatoid arthritis. BMC Musculoskelet Disord. 2013 Jan 8;14:13. doi: 10.1186/1471-2474-14-13. PMID 23294908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in the Asia-Pacific Region from June 2007 to October 2008.
Pre-assignment Details: Screening of subjects occurred up to 2 weeks before randomization followed by a treatment phase of 16 weeks and a 2-week safety follow up.
Groups:
- ETN/MTX: Etanercept (ETN) was administered subcutaneous (SC) bi-weekly (BIW) (eg, on Monday and Thursday, Tuesday and Friday, or Wednesday and Saturday). Each dose of ETN was administered as 1 SC injection.
- DMARD/MTX: Methotrexate (MTX) was taken orally once weekly on the same day of the week (as a single dose or 2 divided doses on the same day) at the same dose subjects were taking at the time of screening. The dose and administration of usual disease-modifying antirheumatic drug (DMARD) therapy followed the approved local label or recommendations. Subjects took commercially available MTX and usual DMARD therapy.
Period: Overall Study
Arm/Group | ETN/MTX | DMARD/MTX
Started | 197 | 103
Completed | 193 | 88
Not Completed | 4 | 15
Not completed — Adverse Event | 3 | 8
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ETN/MTX | DMARD/MTX | Total
Number analyzed (Participants) | 197 | 103 | 300
Age Continuous [Mean (Standard Deviation); unit: years] | 48.38 (11.98) | 48.52 (11.25) | 48.43 (11.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180 | 91 | 271
  Male | 17 | 12 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Adjusted Mean of American College of Rheumatology Response (ACR-N) Area Under Curve (AUC) Over 16 Weeks
Description: ACR-N = the lowest of 3 values (percent change in the number of swollen joints, percent change in the number of tender joints, and median of the other 5 measures in the ACR core data set). Negative numbers indicate worsening.
  The ACR-N AUC was calculated using the trapezoidal rule as the ACR-N multiplied by the duration of the assessment period (in weeks) and was presented as %-weeks.
Time Frame: 16 weeks
Population: The mITT population, defined as all randomly assigned subjects who received at least 1 dose of ETN or MTX in the ETN group or 1 dose of usual DMARD therapy medication or MTX in the usual DMARD therapy group and had at least 1 postbaseline assessment.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | ETN/MTX | DMARD/MTX
Number analyzed (Participants) | 194 | 98
Units on a scale | 434.83 (29.18) | 289.54 (36.11)
Statistical Analysis 1: Comparison: ETN/MTX vs DMARD/MTX; Test type: Superiority or Other; p < 0.001, ANOVA

2. Secondary Outcome: Percentage of Participants Achieving ACR 20, 50, and 70 Responses
Description: Response includes improvement in tender or swollen joints as well as 20 percent improvement in three of the other five criteria. Required: ≥ 20%, 50% or 70% improvement in tender joint count ≥ 20% , 50% or 70% improvement in swollen joint count and at least 20%, 50%, 70% improvement in 3 of the following 5:Patient pain assessment , Patient global assessment ,Physician global assessment, Patient self-assessed disability.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | ETN/MTX | DMARD/MTX
Number analyzed (Participants) | 194 | 98
Percentage of Participants
  ACR 20 | 78.87 | 58.16
  ACR 50 | 56.70 | 34.69
  ACR 70 | 19.07 | 7.14
Statistical Analysis 1: Comparison: ETN/MTX vs DMARD/MTX; ACR 20; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: ETN/MTX vs DMARD/MTX; ACR 50; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 3: Comparison: ETN/MTX vs DMARD/MTX; ACR 70; Test type: Superiority or Other; p = 0.009, Fisher Exact

3. Secondary Outcome: Percentage of Participants Achieving DAS28 <3.2 (Low Disease Activity) and <2.6 (Remission)
Description: Disease Activity Score 28 based on 28 Joints (DAS28) is the calculation of DAS28: DAS28 = 0.56 sqrt (28 painful joint count) + 0.28 sqrt (28 swollen joint count) + 0.70 (ln erythrocyte sedimentation rate (ESR)) + 0.014 (General Health) (GH). GH = Subject general health visual analog scale (0-10 mm).
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | ETN/MTX | DMARD/MTX
Number analyzed (Participants) | 197 | 103
Percentage of Participants
  Low Disease (DAS28 <3.2) | 39.09 | 18.45
  Remission (DAS28 <2.6) | 15.74 | 7.77
Statistical Analysis 1: Comparison: ETN/MTX vs DMARD/MTX; Low Disease (DAS28 <3.2); Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: ETN/MTX vs DMARD/MTX; Remission (DAS28 <2.6); Test type: Superiority or Other; p = 0.069, Fisher Exact

4. Secondary Outcome: Percent Change From Baseline in DAS28 at Week 16
Description: as for outcome 3
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percent change
Arm/Group | ETN/MTX | DMARD/MTX
Number analyzed (Participants) | 197 | 103
Percent change | 38.32 | 27.46
Statistical Analysis 1: Comparison: ETN/MTX vs DMARD/MTX; Test type: Superiority or Other; p < 0.001, ANCOVA

5. Secondary Outcome: Percentage of Participants Achieving European League Against Rheumatism (EULAR) Moderate or Good Response
Description: EULAR Response Criteria DAS28) improvement at week 16. Good response was defined as >1.2 improvement in DAS from Baseline and DAS attained during follow-up of ≤2.4. Non-responders were participants with improvement of ≤0.6 or participants with improvement of >0.6 but ≤1.2 and DAS attained during follow-up of >3.7. Remaining participants were classified as moderate. Scores of good and moderate were considered to have therapeutic response.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | ETN/MTX | DMARD/MTX
Number analyzed (Participants) | 197 | 103
Percentage of Participants | 87.82 | 73.79
Statistical Analysis 1: Comparison: ETN/MTX vs DMARD/MTX; Test type: Superiority or Other; p = 0.003, Fisher Exact

6. Secondary Outcome: Percentage of Participants With DAS28 Improvement of ≥0.6 and ≥1.2
Description: Disease Activity Score 28 based on 28 Joints (DAS28) is the calculation of DAS28: DAS28 = 0.56 sqrt (28 painful joint count) + 0.28 sqrt (28 swollen joint count) + 0.70 (ln erythrocyte sedimentation rate (ESR) + 0.014 (General Health) (GH). GH = Subject general health visual analog scale (0-10 mm).
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | ETN/MTX | DMARD/MTX
Number analyzed (Participants) | 197 | 103
Percentage of Participants
  ≥0.6 | 91.37 | 78.64
  ≥1.2 | 82.74 | 66.02
Statistical Analysis 1: Comparison: ETN/MTX vs DMARD/MTX; ≥0.6; Test type: Superiority or Other; p = 0.003, Fisher Exact
Statistical Analysis 2: Comparison: ETN/MTX vs DMARD/MTX; ≥1.2; Test type: Superiority or Other; p = 0.001, Fisher Exact

7. Secondary Outcome: Percent Change From Baseline in Painful and Swollen Joint Counts
Description: Participant's assessment of pain - A horizontal pain visual analog scale (VAS) (0-100 mm) is used to assess the participants current level of pain; 0 = no pain and 100 = worst pain. Swollen joint count - ACR swollen joint count, an assessment of 28 joints. Joints are classified as either swollen or not swollen.
Time Frame: Week 2, 4, 8, 12, 16
Population: as for outcome 1
Measure: Number; unit: Percent change
Arm/Group | ETN/MTX | DMARD/MTX
Number analyzed (Participants) | 197 | 103
Percent change
  Painful Joints - Week 2 | 34.17 | 27.68
  Painful Joints - Week 4 | 46.11 | 36.71
  Painful Joints - Week 8 | 55.48 | 49.71
  Painful Joints - Week 12 | 65.65 | 55.55
  Painful Joints - Week 16 | 68.99 | 57.31
  Swollen Joints - Week 2 | 38.59 | 21.32
  Swollen Joints - Week 4 | 49.33 | 27.72
  Swollen Joints - Week 8 | 59.91 | 44.19
  Swollen Joints - Week 12 | 67.97 | 50.48
  Swollen Joints - Week 16 | 73.83 | 56.32
Statistical Analysis 1: Comparison: ETN/MTX vs DMARD/MTX; Painful Joints at Week 16; Test type: Superiority or Other; p = 0.014, ANCOVA
Statistical Analysis 2: Comparison: ETN/MTX vs DMARD/MTX; Swollen Joints at Week 16; Test type: Superiority or Other; p < 0.001, ANCOVA

8. Secondary Outcome: Percent Change From Baseline in Physician And Subject Global Assessments
Description: The Physician Global Assessment of Disease Activity: The participant's disease activity is estimated over the last two - three days by the physician; A zero (0) means no disease activity and a ten (10) means extreme disease activity. The Subject Global Assessment of Disease Activity: The participant assesses overall arthritis activity. A zero (0) means no disease activity and a ten (10) means extreme disease activity.
Time Frame: Week 2, 4, 8, 12, 16
Population: as for outcome 1
Measure: Number; unit: Percent change
Arm/Group | ETN/MTX | DMARD/MTX
Number analyzed (Participants) | 197 | 103
Percent change
  Physician Global Assessment - Week 2 | 30.40 | 11.83
  Physician Global Assessment - Week 4 | 39.58 | 22.81
  Physician Global Assessment - Week 8 | 45.86 | 35.41
  Physician Global Assessment - Week 12 | 55.00 | 38.67
  Physician Global Assessment - Week 16 | 62.05 | 45.04
  Subject Global Assessment - Week 2 | 21.84 | 7.24
  Subject Global Assessment - Week 4 | 28.94 | 19.22
  Subject Global Assessment - Week 8 | 34.92 | 26.08
  Subject Global Assessment - Week 12 | 43.18 | 30.10
  Subject Global Assessment - Week 16 | 50.76 | 30.55
Statistical Analysis 1: Comparison: ETN/MTX vs DMARD/MTX; Physician Global Assessment Week 16; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: ETN/MTX vs DMARD/MTX; Subject Global Assessment Week 16; Test type: Superiority or Other; p < 0.001, ANCOVA

9. Secondary Outcome: Percent Change From Baseline in Duration (Minutes) of Morning Stiffness
Description: The duration of morning stiffness on the day of examination should be determined by asking the following two questions: When did you awaken this morning? When were you able to resume your normal activities without stiffness? Duration of morning stiffness is equal to the time elapsed between the above two times in minutes; If none is present enter 0, If morning stiffness is still continuing, please indicate average of duration of stiffness over the past 3 days. If stiffness persists the entire day 1440 minutes (24h x 60 minutes) should be recorded.
Time Frame: Week 2, 4, 8, 12, 16
Population: as for outcome 1
Measure: Number; unit: Percent change
Arm/Group | ETN/MTX | DMARD/MTX
Number analyzed (Participants) | 197 | 103
Percent change
  Week 2 | 54.92 | 16.43
  Week 4 | 63.85 | 33.22
  Week 8 | 73.41 | 37.35
  Week 12 | 79.76 | 52.76
  Week 16 | 80.55 | 46.77
Statistical Analysis 1: Comparison: ETN/MTX vs DMARD/MTX; Week 16; Test type: Superiority or Other; p < 0.001, ANCOVA

10. Secondary Outcome: Percent Change From Baseline in General Health, Pain, and Fatigue, Visual Analog Scales
Description: VAS, participant indicates by marking a vertical line at an appropriate position through a horizontal line. The length of the line measures from left (in mm) and the value (in mm) is recorded. General Health VAS, "in general how would you rate your heath over the last 2-3 weeks", 0mm equals very well and 100mm equals extremely bad. Pain VAS: "indicate the amount of pain experienced during the last 2-3 days", 0 mm equals no pain and 100 mm equals pain as bad as it can be. Fatigue VAS: "how fatigued or tired have you been over the last week", range =No Fatigue - Extremely Fatigued.
Time Frame: Week 2, 4, 8, 12, 16
Population: as for outcome 1
Measure: Number; unit: Percent change
Arm/Group | ETN/MTX | DMARD/MTX
Number analyzed (Participants) | 197 | 103
Percent change
  General Health - Week 2 | 21.14 | 8.88
  General Health - Week 4 | 30.61 | 22.78
  General Health - Week 8 | 38.57 | 27.86
  General Health - Week 12 | 42.10 | 30.26
  General Health - Week 16 | 50.49 | 33.89
  Pain - Week 2 | 27.59 | 9.99
  Pain - Week 4 | 34.73 | 22.98
  Pain - Week 8 | 42.97 | 29.14
  Pain - Week 12 | 48.46 | 33.97
  Pain - Week 16 | 54.42 | 36.45
  Fatigue - Week 2 | 20.90 | 6.63
  Fatigue - Week 4 | 30.87 | 19.00
  Fatigue - Week 8 | 35.92 | 21.82
  Fatigue - Week 12 | 39.65 | 28.65
  Fatigue - Week 16 | 46.92 | 30.04
Statistical Analysis 1: Comparison: ETN/MTX vs DMARD/MTX; General Health Week 16; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: ETN/MTX vs DMARD/MTX; Pain Week 16; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: ETN/MTX vs DMARD/MTX; Fatigue Week 16; Test type: Superiority or Other; p = 0.001, ANCOVA

ADVERSE EVENTS:
Arm/Group | ETN/MTX | DMARD/MTX
Serious Adverse Events (participants affected / at risk) | 6/197 | 3/103
Other Adverse Events (participants affected / at risk) | 66/197 | 71/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ETN/MTX (N=197) | DMARD/MTX (N=103)
Myocardial infarction (Cardiac disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ETN/MTX (N=197) | DMARD/MTX (N=103)
Leukopenia (Blood and lymphatic system disorders) | 4 | 8
Nausea (Gastrointestinal disorders) | 4 | 8
Pyrexia (General disorders) | 6 | 6
Upper respiratory tract infection (Infections and infestations) | 27 | 16
Alanine aminotransferase increased (Investigations) | 11 | 15
Aspartate aminotransferase increased (Investigations) | 7 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.